CLINICAL TRIAL: NCT04626609
Title: Prostaglandin and Cannabinoid Receptors in the Development of Eosinophilic Esophagitis
Brief Title: Prostaglandin and Cannabinoid Receptors in EoE
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: KLI 887-B
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EoE group: Patients with confirmed eosinophilic esophagitis
  Interventions: Other: Biopsy samples; Other: Blood samples
- GERD group: Patients with gastro-esophageal reﬂux disease
  Interventions: Other: Biopsy samples; Other: Blood samples
- Control group: Individuals with no esophageal disease
  Interventions: Other: Biopsy samples; Other: Blood samples

INTERVENTIONS:
Other: Biopsy samples — Esophageal mucosal biopsies are collected during gastroscopy
Other: Blood samples — Blood will be drawn by venipuncture into citrate- or ethylenediaminetetraacetic acid (EDTA)-containing vacutainer tubes and into serum tubes

SUMMARY:
The purpose of this study is to investigate prostaglandin and cannabinoid receptors and their endogenous ligands in eosinophilic esophagitis (EoE). A prostaglandin D2 receptor antagonist has been shown to improve disease symptoms suggesting a regulatory role for bioactive lipids in EoE. Prostaglandin D2 and E2, and endocannabinoids are lipid mediators that govern the functional and inflammatory behavior of immune cells critical for EoE development. The prostaglandin D2 and E2 receptor axis, and the components of the endocannabinoid may be involved in the pathogenesis of EoE.

DETAILED DESCRIPTION:
Prostaglandin D2 and E2 receptors, and components of the endocannabinoid system (cannabinoid receptors and endocannabinoid-metabolizing enzymes) are examined in mucosal esophageal biopsies and blood leukocytes from EoE patients (acute and in remission), individuals with gastroesophageal reflux and from individuals with no esophageal disease. Expression of these components are compared between all cohorts by polymerase chain reaction, Western blots, flow cytometry and immunohistochemical methods. EoE disease activity is evaluated by determining a symptom score and the number of eosinophils per high-power field (hpf) in histologic sections of mucosal biopsies. Additionally, an Endoscopic Reference Score (EREFS) is used. Disease activity is correlated with cannabinoid/prostaglandin D2 and E2 receptor expression. Blood is collected and immediately processed for flow cytometric experiments. Prostaglandins and endocannabinoids are measured in plasma and esophageal mucosal biopsy samples of all cohorts by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed or suspected EoE or GERD
* without esophageal diseases
* with signed informed consent

Exclusion Criteria:

* viral or parasitic diseases (e.g. herpes, candidiasis)
* eosinophilic gastroenteritis, hypereosinophilic syndrome, Crohn's disease
* autoimmune diseases
* unable to give informed consent
* immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing gastroscopy at the outpatients clinic of the Medical University of Graz
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Analysis of cannabinoid receptors- protein content | within 48 months
  Cannabinoid receptors (protein) are measured by flow cytometry in blood leukocytes of patients with EoE (acute and in remission), and of control individuals.
Analysis of cannabinoid receptors- transcripts | within 48 months
  Transcripts of cannabinoid receptors are measured in esophageal mucosal biopsies of patients with EoE (acute and in remission), GERD and in control individuals by polymerase chain reaction.
Analysis of prostaglandin D2 receptors- protein content | within 48 months
  Prostaglandin D2 receptors (protein) are measured by flow cytometry in blood leukocytes of patients with EoE (acute and in remission), and of control individuals.
Analysis of prostaglandin D2 receptors - transcripts | within 48 months
  Transcripts of prostaglandin D2 receptors are measured in esophageal mucosal biopsies of patients with EoE (acute and in remission), GERD and in control individuals by polymerase chain reaction.
Analysis of prostaglandin E2 receptors- protein content | within 48 months
  Prostaglandin E2 receptors (protein) are measured by flow cytometry in blood leukocytes of patients with EoE (acute and in remission), and of control individuals.
Analysis of prostaglandin E2 receptors- transcripts | within 48 months
  Transcripts of prostaglandin E2 receptors are measured in esophageal mucosal biopsies of patients with EoE (acute and in remission), GERD and in control individuals by polymerase chain reaction.

SECONDARY OUTCOMES:
Disease activity Score | within 48 months
  Assessment of a Disease Activity Score:
  The Disease Activity Score will be assessed on the basis of the Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) instrument (Dis Esophagus. 2007;20 (2):130-4) and consists of a questionnaire rated from 0 to 5 where 0 indicates no symptoms while 5 indicates strong symptoms of heartburn and difficulties in swallowing that incapacitates to do daily activities.
Endoscopic Reference Score | within 48 months
  Assessment of an Endoscopic Reference Score:
  Endoscopic findings will be assessed using the EoE Endoscopic Reference Score (EREFS) (Hirano et al. Gut. 2013; 62:489-495) which is composed of 5 classification categories. The classification features include edema, fixed rings, exsudates, furrows and stricture where grade 0 indicates the absence of the feature and grade 2 and 3 increasing severity of the feature.

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Schicho, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No